CLINICAL TRIAL: NCT00603902
Title: A 52-Week, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety and Efficacy of Lorcaserin Hydrochloride in Overweight and Obese Patients
Brief Title: BLOSSOM: Behavioral Modification and Lorcaserin Second Study for Obesity Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APD356-011
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-08

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; lorcaserin; APD356; BLOSSOM; Hypertension; Dyslipidemia; Sleep apnea; glucose tolerance; cardiovascular disease; Arena
MeSH Terms: conditions — Obesity; Weight Loss; Hypertension; Dyslipidemias; Sleep Apnea Syndromes; Cardiovascular Diseases | interventions — lorcaserin; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lorcaserin 10 mg QD (Experimental): Lorcaserin 10 mg tablet each morning and placebo tablet each evening
  Interventions: Drug: Lorcaserin 10 mg once daily (QD)
- Lorcaserin 10 mg BID (Experimental): Lorcaserin 10 mg tablet each morning and evening
  Interventions: Drug: Lorcaserin 10 mg twice a day (BID)
- Matching Placebo (Placebo Comparator): Matching placebo tablet each morning and evening
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Lorcaserin 10 mg once daily (QD) — Lorcaserin 10 mg tablet each morning and placebo tablet each evening for a duration of 52 weeks.
  Other Names: APD356
  Arms: Lorcaserin 10 mg QD
Drug: Lorcaserin 10 mg twice a day (BID) — Lorcaserin 10 mg tablet each morning and evening for a duration of 52 weeks.
  Other Names: APD356
  Arms: Lorcaserin 10 mg BID
Drug: Matching Placebo — Matching placebo tablet each morning and evening for a duration of 52 weeks.
  Arms: Matching Placebo

SUMMARY:
The purpose of this study is to assess the weight loss effect of lorcaserin during and at the end of 1 year of treatment in overweight and obese patients.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group assessment of the effects of lorcaserin hydrochloride during 52 weeks of administration to overweight or obese male and female volunteers aged 18 to 65 years inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and/or obese men and women with a body mass index (BMI) 30 to 45 kg/m2 with or without a comorbid condition (e.g., hypertension, dyslipidemia, CV disease, glucose intolerance, sleep apnea), or 27 to 29.9 kg/m2 with at least one comorbid condition.
* Ability to complete a 1 year study

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus (type I, II or other)
* History of symptomatic heart valve disease
* Serious or unstable current or past medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4008 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arena Pharmaceuticals, Inc., San Diego, California, United States

REFERENCES:
- [Derived] Weissman NJ, Smith SR, Fain R, Hall N, Shanahan WR. Effects of lorcaserin on pre-existing valvulopathy: A pooled analysis of phase 3 trials. Obesity (Silver Spring). 2017 Jan;25(1):39-44. doi: 10.1002/oby.21695. Epub 2016 Nov 26. PMID 27888609
- [Derived] Handelsman Y, Fain R, Wang Z, Li X, Fujioka K, Shanahan W. Lorcaserin treatment allows for decreased number needed to treat for weight and glycemic parameters in week 12 responders with >/=5% weight loss. Postgrad Med. 2016 Nov;128(8):740-746. doi: 10.1080/00325481.2016.1240591. Epub 2016 Oct 19. PMID 27659698
- [Derived] Nguyen CT, Zhou S, Shanahan W, Fain R. Lorcaserin in Obese and Overweight Patients Taking Prohibited Serotonergic Agents: A Retrospective Analysis. Clin Ther. 2016 Jun;38(6):1498-1509. doi: 10.1016/j.clinthera.2016.04.004. Epub 2016 May 17. PMID 27206567
- [Derived] Nesto R, Fain R, Li Y, Shanahan W. Evaluation of lorcaserin on progression of prediabetes to type 2 diabetes and reversion to euglycemia. Postgrad Med. 2016 May;128(4):364-70. doi: 10.1080/00325481.2016.1178590. PMID 27116910
- [Derived] Weissman NJ, Sanchez M, Koch GG, Smith SR, Shanahan WR, Anderson CM. Echocardiographic assessment of cardiac valvular regurgitation with lorcaserin from analysis of 3 phase 3 clinical trials. Circ Cardiovasc Imaging. 2013 Jul;6(4):560-7. doi: 10.1161/CIRCIMAGING.112.000128. Epub 2013 May 9. PMID 23661689
- [Derived] Fidler MC, Sanchez M, Raether B, Weissman NJ, Smith SR, Shanahan WR, Anderson CM; BLOSSOM Clinical Trial Group. A one-year randomized trial of lorcaserin for weight loss in obese and overweight adults: the BLOSSOM trial. J Clin Endocrinol Metab. 2011 Oct;96(10):3067-77. doi: 10.1210/jc.2011-1256. Epub 2011 Jul 27. PMID 21795446
- See also: Arena Pharmaceuticals, Inc. Home Page — http://www.arenapharm.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lorcaserin 10 mg QD: lorcaserin 10 mg once daily (QD) tablets
- Lorcaserin 10 mg BID: lorcaserin 10 mg twice a day (BID) tablets
- Matching Placebo: matching placebo tablets
Period: Overall Study
Arm/Group | Lorcaserin 10 mg QD | Lorcaserin 10 mg BID | Matching Placebo
Started | 802 | 1603 | 1603
Completed | 473 | 917 | 834
Not Completed | 329 | 686 | 769

BASELINE CHARACTERISTICS:
Groups:
- Lorcaserin 10 mg QD: lorcaserin 10 mg QD tablets
- Lorcaserin 10 mg BID: lorcaserin 10 mg BID tablets
- Total: Total of all reporting groups
Arm/Group | Lorcaserin 10 mg QD | Lorcaserin 10 mg BID | Matching Placebo | Total
Number analyzed (Participants) | 801 | 1602 | 1601 | 4004
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.66) | 43.8 (11.81) | 43.7 (11.76) | 43.8 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 656 | 1289 | 1249 | 3194
  Male | 145 | 313 | 352 | 810

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Endpoint- Percentage of Participants Achieving Greater Than or Equal to 5% Weight Loss From Baseline to Week 52
Description: The percentage of patients with a reduction from baseline body weight of 5% or more after 52 weeks.
Time Frame: Baseline and Week 52
Population: Modified Intent to Treat (MITT) with last observation carried forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Lorcaserin 10 mg QD | Lorcaserin 10 mg BID | Matching Placebo
Number analyzed (Participants) | 771 | 1561 | 1541
percentage of participants | 40.2 | 47.2 | 25.0
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Adjustments for baseline body weight; Odds Ratio, log = 2.69, 95% CI 2-sided [2.31 to 3.13]

2. Secondary Outcome: Percent Change in Body Weight From Baseline to Week 52
Description: The percent change in body weight (kg) from baseline to week 52.
Time Frame: Baseline and Week 52
Population: MITT with LOCF
Measure: Least Squares Mean (Standard Error); unit: % change from baseline: body wt (kg)
Arm/Group | Lorcaserin 10 mg QD | Lorcaserin 10 mg BID | Matching Placebo
Number analyzed (Participants) | 771 | 1561 | 1541
% change from baseline: body wt (kg) | -4.75 (0.23) | -5.84 (0.16) | -2.84 (0.16)
Statistical Analysis 1: Comparison: Lorcaserin 10 mg BID vs Matching Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.00, 95% CI 2-sided [-3.44 to -2.56]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Lorcaserin 10 mg QD | Lorcaserin 10 mg BID | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 27/801 | 49/1602 | 36/1601
Other Adverse Events (participants affected / at risk) | 653/801 | 1323/1602 | 1205/1601
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin 10 mg QD (N=801) | Lorcaserin 10 mg BID (N=1602) | Matching Placebo (N=1601)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia facial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Anthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian necrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tethered cord syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Cystocele (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer stage I, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lorcaserin 10 mg QD (N=801) | Lorcaserin 10 mg BID (N=1602) | Matching Placebo (N=1601)
Nausea (Gastrointestinal disorders) | 61 (68) | 145 (160) | 85 (96)
Diarrhoea (Gastrointestinal disorders) | 53 (59) | 98 (119) | 94 (106)
Constipation (Gastrointestinal disorders) | 41 (44) | 80 (91) | 61 (62)
Dry mouth (Gastrointestinal disorders) | 27 (29) | 87 (90) | 37 (41)
Fatigue (General disorders) | 53 (59) | 134 (147) | 66 (71)
Upper respiratory tract infection (Infections and infestations) | 117 (142) | 204 (247) | 202 (238)
Nasopharyngitis (Infections and infestations) | 95 (123) | 201 (240) | 192 (240)
Sinusitis (Infections and infestations) | 67 (77) | 122 (141) | 118 (132)
Urinary tract infection (Infections and infestations) | 61 (80) | 107 (131) | 77 (84)
Back pain (Musculoskeletal and connective tissue disorders) | 55 (60) | 101 (107) | 91 (107)
Headache (Nervous system disorders) | 125 (158) | 250 (293) | 147 (172)
Dizziness (Nervous system disorders) | 50 (58) | 140 (169) | 62 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study results are only allowed with prior written consent from Arena Pharmaceuticals, Inc.